CLINICAL TRIAL: NCT04764513
Title: Safety and Efficiency of γδ T Cell Against Hematological Malignancies After Allo-HSCT. A Dose Escalation, Open-label, Phase 1/2 Study.
Brief Title: Safety and Efficiency of γδ T Cell Against Hematological Malignancies After Allo-HSCT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-062
Record Dates: First submitted 2021-02-19; First posted 2021-02-21 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndromes; Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Lymphoma | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: This dose escalation study will be conducted in two phases. The first phase will have 3 cohorts(Dose escalation, x5 dose increments between cohorts, 2×10^6、 1×10^7/kg and 5×10^7 of cells per kg of body weight). The second phase is an expansion cohort at the maximum tolerated dose determined in the first phase.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with hematological malignancies after allo-HSCT (Experimental): 1. Patients with negative minimal residual disease or stable disease:
     After inclusion, patients will receive or not receive chemotherapy. Subsequently, patients will be dosed with γδ T cell.
  2. Patients with positive minimal residual disease but not hematologic relapse:
     After inclusion, patients will receive chemotherapy. Subsequently, patients will be dosed with γδ T cell.
  3. Patients with hematologic relapse:
  After inclusion, patients will receive chemotherapy. Subsequently, patients will be dosed with γδ T cell.
  Interventions: Biological: Ex-vivo expanded γδ T cell infusion

INTERVENTIONS:
Biological: Ex-vivo expanded γδ T cell infusion — Phase 1: Patients receive ex-vivo expanded γδ T cell (Dose escalation, 3 cohorts, x5 dose increments between cohorts, 2×10^6、 1×10^7 and 5×10^7 of cells per kg of body weight).
  Phase 2: Patients receive ex-vivo expanded γδ T cell at the maximum tolerated dose determined in Phase 1.
  Other Names: Chemotherapy

SUMMARY:
This study investigates the infusion safety and potential curative properties of ex-vivo expanded γδ T cells obtained from the same donor for patients who have hematological malignancies and have accepted allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
This is a single-center, open-label, single-arm study to evaluate the safety and efficacy of ex-vivo expanded γδ T cell in patients with hematological malignancies after allogeneic hematopoietic stem cell transplantation. γδ T cell will be separated from peripheral blood of the same donors. After expansion in vitro, they will be infused to the patients as an immunotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hematological malignancies after allogeneic hematopoietic stem cell transplantation；
2. Age criteria: 18-65 years;
3. Weight criteria: > 40kg;
4. Organ function criteria:

   Cardiac function: Left ventricular ejection fraction (LVEF) ≥40%, Pulmonary function: Indoor oxygen saturation≥95%, Alanine aminotransferase and aspartate aminotransferase ≤ 2.5×ULN (upper limit of normal value), Total bilirubin ≤ 1.5×ULN, Serum creatinine ≤ 1.5×ULN;
5. Life expectancy of at least 4 months;
6. ECOG (Eastern Cooperative Oncology Group) score ≤ 2;
7. Patients able to understand and sign written informed consent.

Exclusion Criteria:

1. GVHD (graft versus host disease) ≥ grade Ⅱ；
2. Thrombotic microangiopathy；
3. Posttransplant lymphoproliferative disorders；
4. Uncontrolled infection or other uncontrolled medical or psychiatric disorders which may preclude patients to undergo clinical studies (discretion of the attending physician)；
5. Patients with chronic diseases that require treatment with immune agents or hormones;
6. Suffering from systemic autoimmune disease or immunodeficiency disease;
7. Systemic use of steroids;
8. Allergic constitution;
9. Hemorrhagic disease or coagulation disorders;
10. Patients participating in other clinical trials within 30 days prior to enrollment;
11. Patients receiving radiotherapy within 4 weeks prior to enrollment;
12. Pregnant or breastfeeding women;
13. According to the researcher's judgment, the patient has other unsuitable conditions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-12 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AEs)[Safety] | Day 28 after completion of treatment
  Safety of γδ T cell assessed by incidence of treatment-emergent adverse events (AEs) per patient graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Incidence of Dose-Limiting Toxicities (DLTs) [Tolerability] | Day 28 after completion of treatment
  Tolerability of γδ T cell assessed by incidence of dose-limiting toxicities (DLTs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Number of patients reaching Complete Remission (CR) [Efficacy] | 12 months post-treatment
  Efficacy of ex-vivo expanded γδ T cell assessed by number of patients reaching Complete Remission (CR).
Overall Survival (OS) [Efficacy] | 12 months post-treatment
  Efficacy of ex-vivo expanded γδ T cell assessed by overall survival (OS) measured in months.
Quality of Life (QoL) | 12 months post-treatment
  Quality of life determined by European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire 'C30'.
Persistence of γδ T cell | Before treatment and up to 3 months after treatment
  Persistence of γδ T cell assessed by number in peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Chunji Gao, Professor, Principal Investigator — Chinese PLA General Hospital; Weidong Han, Professor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China